CLINICAL TRIAL: NCT00564291
Title: Evaluation of Retinal Structure With High Resolution OCT
Brief Title: Evaluation of Retinal Structure With High Resolution Optical Coherence Tomography (OCT)
Status: Completed | Type: Observational
Sponsor: Sebastian Wolf (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Sebastian Wolf, Director, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: KEK 044/07
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Macular Edema; CNV
Keywords: OCT
MeSH Terms: conditions — Macular Edema | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 1: Healthy volunteers
  Interventions: Other: Examination with an OCT device
- 2: CSME secondary to diabetic retinopathy
- 3: ARMD with CNV before and after therapy
  Interventions: Other: Examination with an OCT device
- 4: ARMD atrophic
  Interventions: Other: Examination with an OCT device
- 5: Retinal vein occlusion
  Interventions: Other: Examination with an OCT device
- 6: retinitis pigmentosa
  Interventions: Other: Examination with an OCT device
- 7: vitreoretinal proliferation
  Interventions: Other: Examination with an OCT device

INTERVENTIONS:
Other: Examination with an OCT device
  Groups: 1; 3; 4; 5; 6; 7

SUMMARY:
Comparison of different OCT instruments to assess retinal thickness, correlation to fluorescein angiography, and visual outcome after therapy with anti-VEGF therapy

DETAILED DESCRIPTION:
Comparison of different OCT instruments to assess retinal thickness, correlation to fluorescein angiography, and visual outcome after therapy with anti-VEGF therapy

ELIGIBILITY:
Inclusion Criteria:

* Macular disease
* Healthy subjects

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects and patients with macular diseases
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Integrity of retinal layers | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, MD, PhD, Principal Investigator — University of Bern; Sebastian Wolf, MD PhD, Study Director — University of Bern
Locations (2):
- Switzerland (2):
  - Dep. Ophthalmology, University Hospital Bern, Bern
  - Klinik und Poliklinik für Augenheilkunde, University Bern, Bern

REFERENCES:
- [Derived] Lincke JB, Keller S, Amaral J, Zinkernagel MS, Schuerch K. Ciliary body length revisited by anterior segment optical coherence tomography: implications for safe access to the pars plana for intravitreal injections. Graefes Arch Clin Exp Ophthalmol. 2021 Jun;259(6):1435-1441. doi: 10.1007/s00417-020-04967-3. Epub 2020 Oct 19. PMID 33074373
- [Derived] Wolf-Schnurrbusch UE, Ghanem R, Rothenbuehler SP, Enzmann V, Framme C, Wolf S. Predictors of short-term visual outcome after anti-VEGF therapy of macular edema due to central retinal vein occlusion. Invest Ophthalmol Vis Sci. 2011 May 18;52(6):3334-7. doi: 10.1167/iovs.10-6097. PMID 21087958
- [Derived] Rothenbuehler SP, Waeber D, Brinkmann CK, Wolf S, Wolf-Schnurrbusch UE. Effects of ranibizumab in patients with subfoveal choroidal neovascularization attributable to age-related macular degeneration. Am J Ophthalmol. 2009 May;147(5):831-7. doi: 10.1016/j.ajo.2008.12.005. Epub 2009 Feb 13. PMID 19217019